CLINICAL TRIAL: NCT01998113
Title: Glyburide and Metformin for the Treatment of Gestational Diabetes Mellitus. A Systematic Review and Meta-analysis of Randomized Controlled Trials Comparing These Drugs Either vs Insulin or vs Each Other.
Brief Title: Glyburide and Metformin for the Treatment of Gestational Diabetes Mellitus. Systematic Review
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ADO-2013-153
Record Dates: First submitted 2013-11-08; First posted 2013-11-28 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2013-11

CONDITIONS: Gestational Diabetes Mellitus
Keywords: gestational diabetes mellitus; glyburide; metformin; oral agents; insulin; outcomes
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Glyburide (Glyburide vs Insulin): Glyburide vs Insulin trials
  Interventions: Drug: Glyburide vs Insulin trials
- Insulin (Glyburide vs Insulin): Glyburide vs Insulin trials
  Interventions: Drug: Glyburide vs Insulin trials
- Metformin (Metformin vs Insulin): Metformin vs Insulin trials
  Interventions: Drug: Metformin vs Insulin trials
- Insulin (Metformin vs Insulin): Metformin vs Insulin trials
  Interventions: Drug: Metformin vs Insulin trials
- Metformin (Metformin vs Glyburide): Metformin vs Glyburide trials
  Interventions: Drug: Metformin vs Glyburide trials
- Glyburide (Metformin vs Glyburide): Metformin vs Glyburide trials
  Interventions: Drug: Metformin vs Glyburide trials

INTERVENTIONS:
Drug: Glyburide vs Insulin trials — Affecting groups 1 and 2
  Groups: Glyburide (Glyburide vs Insulin); Insulin (Glyburide vs Insulin)
Drug: Metformin vs Insulin trials — Affecting groups 3 and 4
  Groups: Insulin (Metformin vs Insulin); Metformin (Metformin vs Insulin)
Drug: Metformin vs Glyburide trials — Affecting groups 5 and 6
  Groups: Glyburide (Metformin vs Glyburide); Metformin (Metformin vs Glyburide)

SUMMARY:
Since the publication in the New England Journal of Medicine (NEJM) in 2000 of the Langer's trial comparing glyburide vs insulin in the treatment of gestational diabetes mellitus (GDM), additional studies of oral agents for the treatment of GDM have been published (observational, randomized controlled trials (RCT), and trials using other drugs like metformin).

Some meta-analysis to summarize the evidence have been published: Nicholson 2009 (including 4 RCT addressing different drugs), Dhulkotia 2010 (including 6 RCT addressing different drugs, the meta-analysis combining all drugs altogether), Gui 2013 (including 5 RCT addressing metformin vs insulin).

Oral agents are increasingly used for the treatment of GDM. Investigators aim to update the evidence on RCTs comparing glyburide and metformin vs insulin or between them and summarize this evidence using meta-analysis tools. Specifically, investigators aim at producing distinct meta-analyses for each one of the three drug comparisons. This information is not available in the literature since the most recent systematic reviews specifically dealing on oral agents for the treatment of GDM have addressed a single drug comparison (Gui 2013) or have combined different drug comparisons into a single meta-analysis (Dhulkotia 2010)

DETAILED DESCRIPTION:
This project involves the systematic review of RCT addressing the use of glyburide or metformin for the treatment of GDM. The review will include RCT comparing these drugs versus insulin or making direct comparisons between the two oral agents in pregnant women with GDM.

Investigators have pre-specified a series of maternal and fetal outcomes of interest.

A comprehensive electronic search strategy will be complemented with a search of bibliographies from relevant studies and the contact of authors from the eligible studies regarding issues on study design or information on primary outcomes.

The risk of bias of included studies will be analyzed and this information used to perform sensitivity analyses. If possible, data from original studies will be pooled into relative risks for dichotomous outcomes and mean differences for continuous outcomes.

Heterogeneity will be explored for all the analyses. Analyses will be undertaken using a fixed effects model that will be repeated using a random effects model in case of substantial heterogeneity.

Results of the systematic review will be published following PRISMA guidance.

ELIGIBILITY:
Inclusion Criteria:

* RCT
* GDM
* comparing Glyburide vs Insulin, Metformin vs Insulin or Metformin vs Glyburide
* data on fetal and/or maternal outcomes
* full text available

Exclusion Criteria:

* significant overlap with other articles of the same group

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pregnant women with gestational diabetes mellitus requiring drug treatment
Sampling Method: Probability Sample
Enrollment: 2509 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
3rd trimester glycated hemoglobin | 3rd trimester of pregnancy
  mean difference of 3rd trimester glycated hemoglobin
total maternal weight gain | during pregnancy
  mean difference of total maternal weight gain (as defined by the authors)
severe maternal hypoglycemia | from enrollment to delivery
  relative risk of severe maternal hypoglycemia (as defined by the authors)
preeclampsia | during pregnancy or puerperium
  relative risk of preeclampsia (as defined by the authors)
cesarean section | at the end of pregnancy
  relative risk of cesarean section (as defined by the authors)
gestational age at birth | at birth
  mean difference of gestational age at birth (as defined by the authors)
preterm birth | at birth
  relative risk of preterm birth (as defined by the authors)
birthweight | at birth
  mean difference of birthweight (as defined by the authors)
macrosomia | at birth
  relative risk of macrosomia (defined as birthweight >=4000 g)
large-for-gestational age newborn | at birth
  relative risk of large-for-gestational age newborn (as defined by the authors)
small-for-gestational age newborn | at birth
  relative risk of small-for-gestational age newborn (as defined by the authors)
neonatal hypoglycemia | in the neonatal period
  relative risk of neonatal hypoglycemia (as provided by the authors)
perinatal mortality | in the perinatal period
  relative risk of perinatal mortality (as defined by the authors)
insulin treatment | from enrollment to delivery
  relative risk of insulin treatment (for trials comparing metformin vs glyburide)

SECONDARY OUTCOMES:
fasting blood glucose | in the period from enrollment to delivery
  mean difference of fasting blood glucose (as defined by the authors)
postprandial blood glucose | in the period from enrollment to delivery
  mean difference of postprandial blood glucose (as defined by the authors)
maternal weight gain since enrollment | in the period from enrollment to delivery
  mean difference of maternal weight gain since enrollment (as defined by the authors)
pregnancy-induced hypertension | during pregnancy
  relative risk of pregnancy-induced hypertension (as defined by the authors)
induction of labour | at the end of pregnancy
  relative risk of induction of labour (as described by the authors)
cord C peptide | at birth
  mean difference of cord C peptide (as defined by the authors)
cord insulin | at birth
  mean difference of cord insulin (as defined by the authors)
abnormal 1 min Apgar | at birth
  relative risk of abnormal 1 min Apgar (defined as lower than 7)
abnormal 5 min Apgar | at birth
  relative risk of abnormal 5 min Apgar (defined as lower than 7)
obstetric trauma | at birth
  relative risk of obstetric trauma (as defined by the authors)
severe neonatal hypoglycemia | in the neonatal period
  relative risk of severe neonatal hypoglycemia (as defined by the authors)
neonatal jaundice | in the neonatal period
  relative risk of neonatal jaundice (as defined by the authors)
significant respiratory distress | in the neonatal period
  relative risk of significant respiratory distress (described as respiratory distress syndrome or requiring respiratory support)
stillbirth | in the antenatal period
  relative risk of stillbirth (as defined by the authors)
neonatal mortality | in the neonatal period
  relative risk of neonatal mortality (as defined by the authors)
Neonatal Intensive Care Unit (NICU) admittance | in the neonatal period
  relative risk of NICU admittance (as defined by the authors)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Langer O, Conway DL, Berkus MD, Xenakis EM, Gonzales O. A comparison of glyburide and insulin in women with gestational diabetes mellitus. N Engl J Med. 2000 Oct 19;343(16):1134-8. doi: 10.1056/NEJM200010193431601. PMID 11036118
- [Background] Rowan JA, Hague WM, Gao W, Battin MR, Moore MP; MiG Trial Investigators. Metformin versus insulin for the treatment of gestational diabetes. N Engl J Med. 2008 May 8;358(19):2003-15. doi: 10.1056/NEJMoa0707193. PMID 18463376
- [Background] Dhulkotia JS, Ola B, Fraser R, Farrell T. Oral hypoglycemic agents vs insulin in management of gestational diabetes: a systematic review and metaanalysis. Am J Obstet Gynecol. 2010 Nov;203(5):457.e1-9. doi: 10.1016/j.ajog.2010.06.044. Epub 2010 Aug 24. PMID 20739011
- [Background] Nicholson W, Bolen S, Witkop CT, Neale D, Wilson L, Bass E. Benefits and risks of oral diabetes agents compared with insulin in women with gestational diabetes: a systematic review. Obstet Gynecol. 2009 Jan;113(1):193-205. doi: 10.1097/AOG.0b013e318190a459. PMID 19104375
- [Background] Gui J, Liu Q, Feng L. Metformin vs insulin in the management of gestational diabetes: a meta-analysis. PLoS One. 2013 May 27;8(5):e64585. doi: 10.1371/journal.pone.0064585. Print 2013. PMID 23724063
- [Background] Silva JC, Fachin DR, Coral ML, Bertini AM. Perinatal impact of the use of metformin and glyburide for the treatment of gestational diabetes mellitus. J Perinat Med. 2012 Jan 10;40(3):225-8. doi: 10.1515/jpm-2011-0175. PMID 22505499
- [Derived] Balsells M, Garcia-Patterson A, Sola I, Roque M, Gich I, Corcoy R. Glibenclamide, metformin, and insulin for the treatment of gestational diabetes: a systematic review and meta-analysis. BMJ. 2015 Jan 21;350:h102. doi: 10.1136/bmj.h102. PMID 25609400